CLINICAL TRIAL: NCT01124240
Title: Phase 11 Study of Cilengitide in Combination With Concurrent Chemotherapy and Radiotherapy Followed by Protracted Daily Low Dose Temozolomide and Low Dose Procarbazine D1 - 20 in Newly Diagnosed Glioblastoma Without Methylation of the MGMT Promoter Gene
Brief Title: Temozolomide and Procarbazine With Cilengitide for Patients With Glioblastoma Multiforme Without Methylation of the MGMT Promoter Gene
Acronym: ExCentric
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Sydney and Central Coast Area Health Service (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Dr Helen Wheeler, Royal North Shore Hospital, Sydney, Australia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0910259M
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Newly Diagnosed Non Methylated Glioblastoma Multiforme Grade 4
Keywords: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Cilengitide; Temozolomide; Procarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cilengitide — Cilengitide 2000 mg flat i.v. twice weekly is administered over a period of 18 months without interruption.
  Starting one week after the initiation of Cilengitide, RTX (60 Gy, 2 Gy per fraction) with concurrent daily temozolomide (60 mg/m2 p.o.) and daily procarbazine (PCB, 50 mg p.o. if BSA < 1.7; 100 mg p.o. if BSA ≥ 1.7) is given over a period of 6 weeks (RTX Monday to Friday, both TMZ and PCB seven days a week).
  After a break of 4 weeks, adjuvant TMZ (50mg/m2 p.o in first cycle, 60 mg/m2 p.o. in subsequent cycles) and PCB (50 mg p.o. if BSA < 1.7; 100 mg p.o. if BSA ≥ 1.7) are then given daily D1 to 20. This TMZ/PCB cycle is repeated every 28 days over a total period of 6 cycles.
  Other Names: Temozolomide; Procarbazine

SUMMARY:
Cilengitide 2000 mg flat i.v. twice weekly is administered over a period of 18 months without interruption.

Starting one week after the initiation of Cilengitide, RTX (60 Gy, 2 Gy per fraction) with concurrent daily temozolomide (60 mg/m2 p.o.) and daily procarbazine (PCB, 50 mg p.o. if BSA < 1.7; 100 mg p.o. if BSA ≥ 1.7) is given over a period of 6 weeks (RTX Monday to Friday, both TMZ and PCB seven days a week).

After a break of 4 weeks, adjuvant TMZ (50mg/m2 p.o in first cycle, 60 mg/m2 p.o. in subsequent cycles) and PCB (50 mg p.o. if BSA < 1.7; 100 mg p.o. if BSA ≥ 1.7) are then given daily D1 to 20. This TMZ/PCB cycle is repeated every 28 days over a total period of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed supratentorial GBM (WHO Grade IV,including GBM subtypes, e.g. gliosarcoma), histopathologically confirmed by central assessment as part of the screening for the CENTRIC trial.
2. Males or females ≥18 years of age.
3. Proven unmethylated MGMT gene promoter status, centrally assessed as part of the screening for the CENTRIC trial.
4. Written informed consent for the present trial obtained before undergoing any study-related activities. The informed consent also allows access to all information obtained during the screening for the CENTRIC trial, notably the result of the MGMT testing.
5. Available post-operative Gd-MRI performed within <48 hours after surgery (in case it was not possible to obtain a Gd-MRI within <48 hours post surgery, a Gd-MRI is to be performed prior to randomization).
6. Stable or decreasing dose of steroids for >5 days prior to randomization.
7. ECOG PS of 0-1.
8. Interval of ≥2 weeks but ≤7 weeks after surgery or biopsy before first administration of study treatment.
9. Meets one of the following RPA classifications:

   * Class III (age <50 years and ECOG PS 0).
   * Class IV (meeting one of the following criteria:

     1. Age <50 years and ECOG PS 1 or
     2. Age ≥50 years, underwent prior partial or total tumor resection, Mini Mental State Examination [MMSE]≥27).
   * Class V (meeting one of the following criteria:

     1. Age ≥50 years and underwent prior partial or total tumour resection, MMSE <27 or
     2. Age ≥50 years and underwent prior tumor biopsy only).
10. Laboratory values (within 2 week prior to randomization):

    * Absolute neutrophil count ≥1500/mm3.
    * Platelets ≥ 100,000/mm3.
    * Creatinine ≤1.5 x upper limit of normal (ULN) or creatinine clearance rate ≥60 mL/min
    * Prothrombin time (PT) international normalized ratio (INR) and partial thromboplastin time (PTT) within normal limits.
    * Hemoglobin ≥10 g/dL.
    * Total bilirubin ≤1.5 x the ULN.
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN(except when attributable to anticonvulsants).
    * Alkaline phosphatase ≤ 2.5 x ULN.

Exclusion criteria

Subjects are not eligible for this study, if they fulfill one or more of the following exclusion criteria:

1. Prior chemotherapy within the last 5 years.
2. Prior RTX of the head.
3. Receiving concurrent investigational agents or has received an investigational agent(s) within the past 30 days prior to the first dose of Cilengitide .
4. Prior systemic antiangiogenic therapy.
5. Placement of Gliadel® wafer at surgery.
6. Treatment with a prohibited concomitant medication.
7. Planned surgery for other diseases (e.g. dental extraction).
8. History of recent peptic ulcer disease (endoscopically proven gastric ulcer, duodenal ulcer, or esophageal ulcer) within 6 months of enrollment.
9. History of malignancy. Subjects with curatively treated cervical carcinoma in situ or basal cell carcinoma of the skin, or subjects who have been free of other malignancies for ≥ 5 years are eligible for this study.
10. History of coagulation disorder associated with bleeding or recurrent thrombotic events.
11. Clinically manifest myocardial insufficiency (NYHA III, IV) or history of myocardial infarction during the past 6 months. Uncontrolled arterial hypertension.
12. Concurrent illness, including severe infection, which may jeopardize the ability of the subject to receive the procedures outlined in this protocol with reasonable safety.
13. Subject is pregnant (positive serum beta human chorionic gonadotropin [β-HCG] test at screening) or is currently breast-feeding, anticipates becoming pregnant/ impregnating their partner during the study or within 6 months after study participation, or subject does not agree to follow acceptable methods of birth control, such as hormonal contraception, intra-uterine pessar, condoms or sterilization, to avoid conception during the study and for at least 6 months after receiving the last dose of study treatment.
14. Current alcohol dependence or drug abuse.
15. Known hypersensitivity to the study treatment.
16. Legal incapacity or limited legal capacity.
17. Inability to undergo Gd-MRI.
18. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
19. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or of family members who suffer(ed) from such.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-11 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
12 month progression free survival | 3 years

SECONDARY OUTCOMES:
Objective response | 3 years
  MRI review
Toxicity | 3 years
  Utilising NCI CTC v 3.0
Peripheral WBC MGMT modulation | 3 years
  Blood collection and analysis
biomarker correlation with response | 3 years
  using multiplex bioassay analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Royal North Shore Hospital, Sydney, New South Wales, Australia